CLINICAL TRIAL: NCT00696631
Title: Antiarrhythmic Trial With Dronedarone in Moderate to Severe CHF Evaluating Morbidity Decrease
Brief Title: European Trial of Dronedarone in Moderate to Severe Congestive Heart Failure
Acronym: ANDROMEDA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated as the active treatment was associated with an increased hazard
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC4966; SR33589; NCT00543699 (obsolete NCT alias)
Record Dates: First submitted 2008-06-12; First posted 2008-06-13 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Congestive Heart Failure
Keywords: Heart disease; morbidity
MeSH Terms: conditions — Heart Failure; Heart Diseases | interventions — Dronedarone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dronedarone 400mg bid (Experimental): dronedarone 400mg tablets
  Interventions: Drug: Dronedarone (SR33589)
- Placebo (Placebo Comparator): matching placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronedarone (SR33589) — oral administration
  Other Names: Multaq®
  Arms: Dronedarone 400mg bid
Drug: Placebo — oral administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy, tolerability and safety of dronedarone versus placebo in patients with symptomatic congestive heart failure (CHF) and left ventricular dysfunction (LVD) when added to evidence based treatments for CHF.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized with symptomatic CHF, current New York Heart Association (NYHA) class II-IV requiring treatment with a diuretic, who had had within the last month at least 1 episode of dyspnea or fatigue at rest, or on slight exertion corresponding to NYHA class III or IV
* Wall motion index (WMI) ≤1.2 determined by a blinded central evaluation of a recorded standard echocardiography, equivalent to a left ventricular ejection fraction (LVEF) ≤35%.

Exclusion Criteria:

* acute pulmonary edema within 12 hours prior to start of study medication
* various heart conditions (cardiogenic shock, obstructive valvular disease, obstructive cardiomyopathy; acute myocardial infarction, cardiac surgery, acute myocarditis or constrictive pericarditis, history of torsades de pointes, bradycardia <50 bpm and/or PR-interval ≥280 ms, QTc-interval >500 ms, significant sinus node disease)
* any illness or disorder other than CHF (cancer with metastasis, organ transplantation)
* current participation in another clinical study or currently taking an investigational drug including dronedarone or concomitant prohibited medication or treatment with other class I or III anti-arrhythmic drugs
* pregnant and/or breastfeeding women or women of child-bearing potential without adequate birth control
* serum potassium <3.5 mmol/L.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 653 (Actual)
Dates: Start 2002-06; Primary Completion 2003-01 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Death from any cause or adjudicated hospitalization for worsening heart failure | Until study cut-off date

CONTACTS AND LOCATIONS:
Overall Officials: ICD, Study Director — Sanofi
Locations (6):
- Sanofi-aventis Administrative Office, Hørsholm, Denmark
- Sanofi-aventis Administrative Office, Budapest, Hungary
- Sanofi-aventis Administrative Office, Gouda, Netherlands
- Sanofi-aventis Administrative Office, Lysaker, Norway
- Sanofi-aventis Administrative Office, Warsaw, Poland
- Sanofi-aventis Administrative Office, Bromma, Sweden

REFERENCES:
- [Result] Kober L, Torp-Pedersen C, McMurray JJ, Gotzsche O, Levy S, Crijns H, Amlie J, Carlsen J; Dronedarone Study Group. Increased mortality after dronedarone therapy for severe heart failure. N Engl J Med. 2008 Jun 19;358(25):2678-87. doi: 10.1056/NEJMoa0800456. PMID 18565860